CLINICAL TRIAL: NCT02226042
Title: Investigating the Neuropsychological Mechanisms Underlying Mindfulness-based Cognitive Therapy
Brief Title: Investigating the Mechanisms of Mindfulness-based Cognitive Therapy (MBCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Kate Williams, PhD Student, University of Manchester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MBCTMechanisms
Record Dates: First submitted 2014-08-21; First posted 2014-08-26 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Major Depression (in Remission)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness-based Cognitive Therapy (Experimental): Individuals currently in remission from depression will choose to enter the Mindfulness-based Cognitive Therapy (MBCT) arm and undergo the 8 week MBCT group programme
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy
- Non-MBCT arm (No Intervention): Individuals currently in remission from depression will choose not to undergo the 8 week MBCT group programme
- Healthy volunteers (No Intervention): Individuals who have never experienced major depression

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy — MBCT: Mindfulness-based Cognitive Therapy is an 8 week group-based programme consisting of approximately 12 participants per group. There is also a full one day of practice around week 6. MBCT was initially designed for individuals in remission from depression and at risk of relapsing. The intervention is a mix of mindfulness meditation, cognitive behavioural therapy exercises and psychoeducation. MBCT has been shown to be effective in reducing relapse risk over 12 months.
  Other Names: MBCT
  Arms: Mindfulness-based Cognitive Therapy

SUMMARY:
This research will investigate the neuropsychological mechanisms underlying the eight-week Mindfulness-based Cognitive Therapy (MBCT) programme.

Participants in remission from depression will be seen pre- and post-MBCT to assess the underlying neuropsychological mechanisms. All will be followed-up over 12 months to assess the relationship of these neuropsychological changes with relapse risk.

The research will focus primarily on changes in self-compassion, rumination, attention and structural brain changes, with secondary focus on other mechanisms of emotional processing and memory.

DETAILED DESCRIPTION:
There will be three groups in total.

* The first group will take 36 participants in remission from major depression (rMDD) through the 8 week MBCT program.
* A control group of 36 rMDD participants will not receive the intervention.
* A group of never depressed healthy control participants will also be recruited.

Research visits for participants not undergoing MBCT will be separated by an 8 week gap.

All participants will be seen before and after the 8 weeks for completion of neuropsychological assessments and questionnaires.

rMDD participants will be followed up over the following 12 months to identify any predictors of relapse.

ELIGIBILITY:
Inclusion Criteria:

Participants with remitted depression (rMDD):

* At least two previous episodes of DSM-IV major depression in adulthood, diagnosed using the Mini International Neuropsychiatric Interview (M.I.N.I).
* Full or partial remission for at least three months with two depressive episodes within the last five years.
* A score of less than or equal to 12 on the Montgomery Asberg Depression Rating Scale (MADRS) mood assessment.
* If on medication, no recent or planned major changes

Healthy volunteers:

* In good psychological health screened with the M.I.N.I

All participants:

* in good physical health (to reduce risk of confounding physical health problems).
* sufficiently fluent in English to ensure valid understanding and completion of the tasks.
* minimum I.Q level of 80 to ensure sufficient understanding of the neurocognitive tasks administered.
* colour vision and acuity within normal/corrected to normal limits.

Exclusion criteria:

* Any current mental health diagnosis (DSM-IV diagnosis including current major depression, bipolar disorder, psychosis, Obsessive Compulsive Disorder (OCD), substance abuse or dependence, eating disorders)
* Physical health or neurological disorders that might interfere with the interpretation of the tasks, including a history of significant head injury.
* In addition healthy volunteers will be without a history mental health disorders (DSM-IV)
* Current or previous experience of mindfulness-based treatments or extensive cognitive behavioural treatment, or planned participation in psychological treatments during the key time for the study (between pre and post visits).
* Planned major alteration in drug treatment for depression between pre and post visits.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Changes in self-compassion following MBCT measured by both neuropsychological and self-report measures | measured at baseline and post intervention (8 weeks post baseline) and at each follow-up visit (3 in total)
  Two neuropsychological measures of self-compassion have been developed and will be administerat baseline and after MBCT/8 week gap (8 weeks post baseline). Self-report questionnaires will be administered before and after MBCT/8 week gap and at subsequent follow-up visits (3, 6, 12 months).

SECONDARY OUTCOMES:
Changes in levels of rumination following MBCT measured through both neuropsychological and self-report measures | measured at baseline and after the intervention/8 week gap (8 weeks post baseline) and at each follow-up visit (3 in total)
  One neuropsychological measure of rumination has been developed and will be administered at baseline and immediately after MBCT/8 week gap (8 weeks post baseline).
  Self-report questionnaires will be administered at baseline and after MBCT/8 week gap (8 weeks post baseline) and at subsequent follow-up visits (3,6,12 months).
Changes in attention regulation following MBCT | measured at baseline and after the intervention/8 week gap (8 weeks post baseline)
Changes in brain structure following MBCT | measured at baseline and after the intervention (8 weeks post baseline)

OTHER OUTCOMES:
Changes in emotional processing | measured at baseline and after the intervention/8 week gap (8 weeks post baseline)
  Other neuropsychological assessments of emotional processing (face emotion recognition, memory, cognitive flexibility) will be assessed at baseline and after MBCT/8 week gap (8 weeks post baseline).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams K, Hartley S, Anderson IM, Birtwell K, Dowson M, Elliott R, Taylor P. An ongoing process of reconnection: A qualitative exploration of mindfulness-based cognitive therapy for adults in remission from depression. Psychol Psychother. 2022 Mar;95(1):173-190. doi: 10.1111/papt.12357. Epub 2021 Jul 17. PMID 34272797